CLINICAL TRIAL: NCT00393185
Title: Non-myeloablative Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Primary Biliary Cirrhosis: A Phase I Study
Brief Title: Stem Cell Transplantation in Patients With Primary Biliary Cirrhosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Burt, MD (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Immunosuppression; Primary Biliary Cirrhosis; Allogeneic Hematopoietic Stem Cell
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Non-myeloablative Hematopoietic Stem Cell Transplantation — autologous Hematopoietic Stem Cell Transplantation

SUMMARY:
This disease is believed to be due to immune cells, cells which normally protect the body, but are now destroying the bile ducts in the liver. When the ducts are damaged, bile builds up in the liver and damages liver tissue. Over time, the disease can cause cirrhosis and may make the liver stop working. This study is designed to examine whether treating patients with high dose Cyclophosphamide and Fludarabine (drugs which reduce the function of your immune system) and CAMPATH-1H (a protein that kills the immune cells that are thought to be causing PBC), followed by return of blood stem cells that have been previously collected from patient brother or sister will stop or reverse the disease. The purpose of the Cyclophosphamide, Fludarabine and CAMPATH-1H is to decrease immune system. The purpose of the stem cell infusion is to restore blood production, which will be severely impaired by the Cyclophosphamide, Fludarabine and CAMPATH-1H, and to produce a normal immune system that will no longer attack the body.

DETAILED DESCRIPTION:
There will be no randomization in this study. All subjects who are determined to be eligible for the study treatment will receive high dose cyclophosphamide, fludarabine and CAMPATH-1H followed by infusion of allogeneic peripheral blood stem cells. The procedures the subject will undergo are as follows:

1. Physician visit to determine potential eligibility for the study. Subjects will be evaluated by a transplant physician. They will have a complete physical examination and will provide a full medical history at these visits. In addition, subjects will be asked to complete a quality of life Questionnaire . Finally, the study will be described in detail by the transplant physician and nurse and the consent form will be provided to be taken home to read.
2. HLA Testing. In order to proceed on this study, subjects will need to have a HLA identical matched sibling donor. The subject and his or her siblings will need to undergo HLA typing in order to determine whether there is a match or Cord blood stem cells will be obtained from the New York Blood Center Cord Blood Registry which is an internationally recognized registry or, if a match is not available, from Stemcyte, a commercial registry that specializes in minority donors. One unit of HLA matched cord blood unit will be infused on day zero.
3. Insurance verification. Subjects who remain interested in pursuing the study treatment and who have severe scleroderma that is following a progressive course will proceed to the insurance verification phase. Third party payment or self-pay must be verified before subjects can proceed.
4. Consent form. Prior to proceeding, the appropriate signatures will be obtained on the consent form. Subjects will be given an opportunity to ask further questions of the attending physician and transplant nurse prior to signing the consent form.
5. Pre-transplant testing. To determine final eligibility for the study, subjects will undergo a series of tests/procedures. These include: CXR, electrocardiogram, endoscopy , ultrasound of the liver and gallbladder,transvenous liver biopsy, lymphopheresis, pulmonary function test, urinalysis, and blood testing to include CBC; chemistries; liver and kidney function tests; PT; PTT; AMA; viral studies and, for females, a pregnancy test. Subjects will also be evaluated by a dentist at Northwestern Memorial Hospital to rule out any potential sources of infection. All pre-transplant testing is routine medical testing done to verify diagnosis and to insure adequate organ function and absence of viral illnesses which would preclude a safe transplant course. Allogeneic donors will also need to undergo testing in order to determine eligibility to proceed. Testing for donors will include history and physical, electrocardiogram, CXR, urinalysis, CBC, chemistries, PT, PTT, viral studies and, for females, a pregnancy test.
6. Allogeneic peripheral blood stem cell collection. Allogeneic donors will undergo a routine procedure for the mobilization and collection of peripheral blood stem cells. This includes the subcutaneous administration of G-CSF, to be self-administered as an outpatient, beginning three days prior to the start of peripheral blood stem cell harvesting. The peripheral blood stem cells will be collected as an outpatient in the Blood Center on the fourth day of G-CSF administration. A central line may be placed for this purpose on the first day of leukopheresis. Leukopheresis will be continued on a daily basis (up to four consecutive days) until an adequate number of peripheral blood stem cells have been collected. G-CSF will continue to be administered until leukopheresis is completed. The pheresis catheter will be discontinued when stem cell harvesting is completed. Processed cells will be frozen and stored until they are reinfused after the conditioning regimen.
7. Study treatment. Prior to the administration of the study treatment, subjects will have a double lumen PICC line placed for the administration of chemotherapy, IV fluids, blood products and the withdrawal of blood samples. The placement of a central catheter is a routine medical procedure. Subjects will then undergo conditioning which will include 4 days of intravenous fludarabine and 4 days of cyclophosphamide and 2 days of CAMPATH-1H. All drugs are FDA approved drugs. The previously collected allogeneic peripheral blood stem cells will be reinfused following the completion of the conditioning regimen.
8. Post-transplant follow-up. Subjects will have a history and physical by the transplant physician at 6 months, 12 months, and yearly for 5 years. In addition, routine urinalysis and blood testing will be performed at these same intervals to include CBC; chemistries; kidney and liver function tests; AMA; ultrasound of the liver and gallbladder, transvenous liver biopsy, lymphopheresis, and patients will also be asked to complete a SF-36 Questionnaire, NDDK-QA Questionnaire.

ELIGIBILITY:
Patient enrollment

Inclusion Criteria:

* Age > 55 years old at the time of evaluation
* An established diagnosis of PBC, i.e. presence of all three diagnostic criteria, detectable serum AMA at titer >1:40, elevated alkaline phosphatase levels for > 6 months, and compatible liver histology
* Incomplete response to UDCA at 13-15 mg/kg/day (Incomplete response is defined as elevated serum alkaline phosphatase (>2X upper normal value) after 12 months of UDCA therapy, as defined by Angulo and colleagues).

And any of the following

* Pruritus unresponsive to medical therapy
* Liver disease with more than 50% probability of dying or needing a LTx in the following 36 months according to the Mayo survival model(equivalent to a Mayo score higher than 6.78 (The Mayo survival model is a validated survival instrument based on age, bilirubin PT, and edema that does not require a liver biopsy).

Exclusion Criteria:

* Poor performance status (ECOG > 2) at the time of entry
* Serum bilirubin > 4.0 mg/dl
* Significant end organ damage such as:

  1. LVEF < 40% or deterioration of LVEF during exercise test on MUGA or echocardiogram
  2. Untreated life-threatening arrhythmia
  3. Active ischemic heart disease or heart failure
  4. End-stage lung disease characterized by DLCOadj < 45% of predicted value
  5. Serum creatinine > 2.0 mg/dl
* HIV positive
* Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment
* Prior history of malignancy except localized basal cell or squamous skin cancer; Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis
* Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
* Inability to give informed consent
* Major hematological abnormalities such as platelet count < 100,000/ul or ANC < 1000/ul
* GI bleed from portal hypertension
* Portal HTN documented by transvenous portal vein wedge pressure greater than 20 cm H20
* Ascites that is non-responsive to full-dose diuretics and human albumin infusion
* Systemic sclerosis
* AMA positive donor
* HCV PCR positive or HBSAg positive donor
* Failure to collect less than 2.0 x 106 CD34 cells/kg from a matched sibling
* Patient on liver transplant list

Donor enrollment

Inclusion Criteria:

* Donor must be a HLA identical sibling or HLA matched cord blood donor.
* If multiple HLA matched donors are available, preference will be given to same sex, same CMV status, or in the case of cord blood higher nucleated cell count.
* AMA negative
* If no HLA matched sibling is available, donor may be HLA matched cord blood. The minimum number of cord blood nucleated cells available must be more than 2X107/kg. To achieve this number of nucleated cells, two units of HLA matched cord blood may be utilized (Wagner JE Blood 2005 Feb 1; 105(3): 1343-7)

Exclusion criteria:

* Physiologic age > 50 years old or <18 years old (except cord blood units)
* HIV positive
* Active ischemic heart disease or heart failure
* Acute or chronic active hepatitis
* Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the donor to tolerate stem cell collection
* Prior history of malignancy except localized basal cell or squamous skin cancer; Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis
* Positive pregnancy test
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
* Major hematological abnormalities such as platelet count less than 100,000/ul, ANC less than 1000/ul

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
No liver-related death or LTx over the 2-year (extended to 5 years) follow-up; Normalization of serum alkaline phosphatase over 6 months;Amelioration of PBC histological stage with reduction of both inflammation and fibrosis scores 42 | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University